CLINICAL TRIAL: NCT00000889
Title: A Randomized, Open-Label, Phase II Study of Subcutaneous Interleukin-2 (Proleukin) Plus Antiretroviral Therapy vs. Antiretroviral Therapy Alone in Patients With HIV Infection and at Least 350 CD4+ Cells/mm3
Brief Title: A Study to Evaluate the Effects of Giving Interleukin-2 (IL-2) Plus Anti-HIV Therapy to HIV-Positive Patients With CD4 Cell Counts of at Least 350 Cells/mm3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: IRP 021A; 10467 (Registry Identifier: DAIDS ES); SQ 1 ARG; SQIL-2 Argentina
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Interleukin-2; CD4 Lymphocyte Count; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — aldesleukin

INTERVENTIONS:
Drug: Aldesleukin

SUMMARY:
To demonstrate the safety and tolerability of subcutaneously administered interleukin-2 (IL-2) plus antiretrovirals in patients with HIV infection and CD4 counts of 350 cells/mm3 or more. To demonstrate the immunological efficacy of subcutaneous IL-2 therapy plus antiretroviral therapy relative to antiretroviral therapy alone.

IL-2, given through injection under the skin, in combination with anti-HIV therapy can increase CD4 cell counts. This study examines 3 doses of IL-2 in order to determine the safest and most effective dose to use.

DETAILED DESCRIPTION:
Interleukin-2 administered subcutaneously, in combination with antiretrovirals, results in increases in CD4+ cell count that might impact upon HIV disease progression. A Phase III trial involving large numbers of HIV-positive patients is the next step in the development process. To develop appropriate clinical experience with the combination, this Phase II trial will allow administration of IL-2 plus antiretroviral therapy to a small number of patients in sites being considered for the Phase III trial.

Patients are randomized to control therapy with antiretrovirals alone (36 patients) or antiretrovirals plus IL-2 given subcutaneously every 12 hours for 5 days every 8 weeks. Three doses of IL-2 are studied, with 12 patients evaluated at each dose.

If at least 9 of the first 12 patients complete the 5-day dosing period without dose-limiting toxicities, the next 12 patients randomized are treated with the next higher dose; if this dose is tolerated, the last 12 patients randomized receive the highest study dose. Patients enrolled at the first two doses of IL-2 who complete three courses have their dose escalated to a maximum of the highest dose.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a CD4 cell count greater than or equal to 300 cells/mm3.
* Are at least 18.
* Have been on antiretroviral therapy for at least 7 days prior to study entry.

Exclusion Criteria

You will not be eligible for this study if you:

* Abuse alcohol or drugs, or have any serious psychiatric or medical illnesses that would affect your safety or ability to complete the study.
* Have a history of cancer (other than Kaposi's sarcoma), an AIDS-defining illness, a central nervous system (CNS) abnormality, or an autoimmune/inflammatory disease.
* Are pregnant or breast-feeding.
* Have ever received IL-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 1997-10; Primary Completion 1999-12 (Actual); Study Completion 1999-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Losso, Study Chair
Locations (4):
- Argentina (4):
  - Hospital de Clinicas 'Jose de San Martin' C601-040 CRS, Ciudad de Buenos Aires, Buenos Aires
  - Hospital F.J. Muniz C601-050 CRS, Ciudad de Buenos Aires, Buenos Aires
  - Hospital General de Agudos J.M. Ramos Mejia CPCRA CRS, Ciudad de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires C601-020 CRS, Ciudad de Buenos Aires, Buenos Aires